CLINICAL TRIAL: NCT05252689
Title: Clinical Evaluation of Teeth Prepared With Vertical Preparation Technique Versus Deep Chamfer for Monolithic Zirconia Crowns
Brief Title: Clinical Evaluation of Teeth Prepared With Vertical Preparation Versus Deep Chamfer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mai Salah Ibrahim Afifi Elgohary, Assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEBD-CU-2019-9-2
Record Dates: First submitted 2022-02-14; First posted 2022-02-23 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Single Posterior Crowns; Endodontically Treated Teeth; Decayed Teeth
MeSH Terms: conditions — Tooth, Nonvital; Dental Caries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- monolithic zirconia single posterior crowns with deep chamfer finish line (Active Comparator): monolithic zirconia single posterior crowns with deep chamfer finish line fabricated by cad cam machine and cemented by self adhesive resin cement.
  Interventions: Other: monolithic zirconia single posterior crowns with deep chamfer finish line
- monolithic zirconia single posterior crowns with vertical finish line (Experimental): monolithic zirconia single posterior crowns with vertical finish line fabricated by cad cam machine and cemented by self adhesive resin cement.
  Interventions: Other: monolithic zirconia single posterior crowns with vertical finish line

INTERVENTIONS:
Other: monolithic zirconia single posterior crowns with deep chamfer finish line — deep chamfer of 1 mm average thickness for cervical finish line, a convergence angle of 6-12° on each side and up to 20° total, in some studies, is acceptable and occlusal reduction of 1,5-2 mm
  Arms: monolithic zirconia single posterior crowns with deep chamfer finish line
Other: monolithic zirconia single posterior crowns with vertical finish line — using special round-ended 2 degrees tapered diamond burs a non-working tip (batt bur). It has coronal diameter of 1.2 mm, apical diameter of 0.7 mm, and non- cutting end of 1 mm, which reduces or avoids damage to the connective attachment and allows a tooth-guided preparation procedure
  Arms: monolithic zirconia single posterior crowns with vertical finish line

SUMMARY:
It has been demonstrated that a great amount of tooth structure is lost during the prosthetic preparations of abutments for full-coverage FDPs with tooth substance removal of 63% of 73%, this aggressive loss of tooth structure usually accompanied with pain and post-operative sensitivity. In comparison with the vertical preparation technique, there is less amount of tooth substance loss. this clinical study will provide benefits for practitioners and clinicians by guiding them to choose a more conservative treatment plan with the better marginal fit, clinical performance and satisfaction for the patients on the long term. rather than other benefits like less chair time, less risk for pulp injury, less time and cost

DETAILED DESCRIPTION:
A healthy relationship between dental restorations and the periodontium is of prime importance for the clinical longevity and esthetic harmony of full coverage restorations . One of the Most Common complications, derived from fixed prostheses is gingival recession, which constitutes an important clinical concern. This problem is largely associated with iatrogenic effects produced during dental preparation or as a result of poor prosthetic fit which can cause chronic inflammation leading to gingival margin recession around the restoration .

ELIGIBILITY:
Inclusion Criteria:

1. The patients in this study will be in the range of 18-50 years
2. Have no active periodontal or pulpal diseases, have teeth with good restorations
3. Psychologically and physically able to withstand conventional dental procedures
4. Able to return for follow-up examinations and evaluation
5. No tooth mobility or grade 1 can be accepted
6. Patients with teeth problems indicated for single posterior crowns:

   1. Badly decayed teeth
   2. Teeth restored with large filling restorations
   3. Endodontically treated teeth
   4. Malformed teeth
   5. Malposed teeth (Tilted, over-erupted, rotated, etc.)
   6. Spacing between posterior teeth

Exclusion Criteria:

1. Patients under the age of 18 or being incapable of taking out a contract
2. Patient with active resistant periodontal diseases
3. Patients with any medical condition that impaired correct oral hygiene
4. a conspicuous medical or psychological history
5. bruxism, or known allergic reaction to the materials used.
6. pregnant female patients

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Marginal adaptation | 1 year
  Assessed using the modified usphs criteria by Discrete (scores) Alpha (A) No visible evidences of crevice along the margins; no catch or penetration of the explorer.
  Bravo (B) Visible evidence of crevice and/or catch of explorer; no penetration of the explorer.
  Charlie (C) Visible evidence of crevice and penetration of the explorer.

SECONDARY OUTCOMES:
Fracture of the restoration | 1 year
  Assessed using the modified usphs criteria by Discrete (scores) Alpha (A) Smooth surface of the restoration (shiny after air drying)
  Bravo (B) Dull surface and/or chipping of porcelain that does not impair function
  Charlie (C) Chipping of veneering material impairing esthetics and function and/or exposing framework material
gingival inflammation | 1 year
  Assessed using the modified usphs criteria by Discrete (scores) Alpha (A) Normal gingiva
  Bravo (B) Mild inflammation - slight change in color and slight edema but no bleeding on probing;
  Charlie (C) Moderate inflammation redness, edema, and glazing, bleeding on probing;
Recurrent caries | 1 year
  Assessed using the modified usphs criteria by Discrete (scores) Alpha (A) No caries present Bravo (B) Caries present

OTHER OUTCOMES:
Patient satisfaction | 1 year
  VAS (Questionnaire) by Numerical (discrete) ("0" unsatisfied - "10" satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Maha Taymour, PhD, Study Director — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No